CLINICAL TRIAL: NCT04955353
Title: A Double-blind, Randomized, Placebo-controlled Trial to Evaluate the Efficacy of a Hydrolyzed Chicken Collagen Type II Supplement in Alleviating Joint Discomfort
Brief Title: Efficacy of a Hydrolyzed Chicken Collagen Type II in Alleviating Joint Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avicenna Nutraceutical (Other)
Collaborators: BioScreen Testing Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BCS 17-033
Record Dates: First submitted 2021-06-16; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Joint Discomfort

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVC-H2 (Experimental): Participants received Avicenna Hydrolyzed Chicken Collagen Type II (AVC-H2), 2.5g daily, for 8 weeks.
  Interventions: Dietary Supplement: AVC-H2
- Placebo (Placebo Comparator): Participants received placebo of matching amount to that of AVC-H2 daily for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AVC-H2 — A total of 2.5g AVC-H2 daily (2 tablets in the morning and 2 in the evening)
  Arms: AVC-H2
Dietary Supplement: Placebo — A total of 2.5g placebo daily (2 tablets in the morning and 2 in the evening)
  Arms: Placebo

SUMMARY:
Joint pain and disease affect more than one in four adults in the United States. We conducted a double-blind, randomized, placebo-controlled trial to investigate the efficacy of a hydrolyzed chicken collagen type II (HCII) supplement in reducing joint-related discomfort such as pain and stiffness, and in improving mobility. We enrolled adults aged 40-65y (65.5% were women) who had joint discomfort, but had no co-morbidities, and were not taking pain medications. The participants were randomized to receive either the HCII supplement (n=47) or a placebo (n=43) for eight weeks. At baseline, week 4, and week 8, we administered the Western Ontario and McMaster Universities Arthritis Index (WOMAC) survey with three additional wrist-related questions and the Visual Analog Scale for assessments of joint-related symptoms.

DETAILED DESCRIPTION:
Joint pain and disease affects more than one in four adults in the United States. Hydrolyzed Chicken Collagen Type II, hereinafter referred to as HCII, may repair or regenerate deteriorating collagen, and therefore, help address the underlying cause of joint discomfort. This study evaluated the efficacy of Avicenna's patented Hydrolyzed Chicken Collagen Type II product, hereinafter referred to as AVC-H2, in the reduction of joint pain & stiffness and improvement in joint function.

BioScreen Clinical Services conducted a double-blind, randomized, placebo-controlled trial. 90 participants were enrolled, 47 in the AVC-H2 group and 43 in the placebo group; aged 40-65 with overall joint discomfort but no co-morbidities were enrolled. Participants in both groups took two pills in the morning and evening for 8 weeks. The Western Ontario and McMaster Universities Arthritis Index (WOMAC) survey with the addition of 3 questions pertaining to the wrist and Visual Analog Scale (VAS) for pain assessment were conducted at baseline, week 4, and week 8.

The product used was Avicenna's Hydrolyzed Chicken Collagen Type II raw material product. The techniques used to create AVC-H2 mimic the body's natural hydrolysis process for ease of digestion and optimum low molecular weight. AVC-H2 protein consists of protein bonds that have been broken down or "untied" so that they are more easily absorbed by the small intestines. The total collagen in the product is ≥ 70%, making it a highly pure product, in comparison to other collagen products that were tested prior to the study. Total collagen content of AVC-H2 was based off of certificates of analyses prior to the study. As such, a smaller dosage was administered to participants compared to previous studies of similar products. Participants in the study were randomly assigned to receive either 2.5g of AVC-H2 daily or a matching amount of placebo.

Intent to Treat Analysis and Sensitivity Analysis were both used. Intent to Treat Analysis included all study participants and Sensitivity Analysis removed participants who broke protocol and those who initially claimed they had 0 joint pain & stiffness.

To the investigators' knowledge, Avicenna's study appears to be the first to assess the efficacy of HCII on joint discomfort in the wrist and in individuals not taking additional pain medications.

ELIGIBILITY:
Inclusion Criteria:

* men and women 40-65 years of age
* all races
* good general health (free of any systemic or dermatological disorder) but have joint pain, stiffness, or other joint-related discomfort
* literate and able to understand the informed consent document, as well as able to choose whether or not to sign the form
* able to complete a preliminary medical history, Health Insurance Portability and Accountability Act (HIPAA), and Code of Conduct form
* able to cooperate with the Investigator and research staff
* willing and able to comply with the instructions to use the test product, and to complete the full course of the study
* agree to not participate in any other study during the entire duration of the study
* have not participated in a similar study in the past thirty days
* agree to refrain from using any joint-pain relief products except for the product received from our re-search staff during the entire duration of the study
* agree to take a urine pregnancy test prior to enrollment

Exclusion Criteria:

* individuals currently taking any medications that may mask or interfere with the test results
* those who had a history of any acute or chronic disease that would interfere with or increase the risk of study participation
* those with a history of diseases of chronic inflammation (e.g., septic arthritis, gout, and rheumatoid arthritis)
* those who had a recent injury in the hip, knee, and/or wrist in the past six months
* those who had a history of hip, knee, and/or wrist surgery
* those who had injections to reduce joint discomfort in the past 12 months
* those who are at high risk of adverse outcomes for participating in the study and thus may invalidate the study due to confounding factors
* pregnancy or lactation
* individuals who had diabetes or hyperuricemia
* body mass index > 30 kg/m2
* history of substance abuse
* known history of hypersensitivity to any cosmetics, personal care products, or fragrances
* known allergy to eggs, chicken, or any other ingredients in the test product
* individuals who have phenylketonuria
* those who need to take calcium supplementation
* those who are affiliated with the clinical trial agency

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) - Baseline | Baseline
  The WOMAC survey is used to assess joint-related discomfort at baseline. Our version of WOMAC score (adding up from all domains) can range from 0 (min) to 108 (max). The lower the number, the better the outcome (less joint-related discomfort).
Western Ontario and McMaster Universities Arthritis Index (WOMAC) - Midpoint (Week 4) | Week 4
  The WOMAC survey is used to assess joint-related discomfort at midpoint of the study. Our version of WOMAC score (adding up from all domains) can range from 0 (min) to 108 (max). The lower the number, the better the outcome (less joint-related discomfort).
Western Ontario and McMaster Universities Arthritis Index (WOMAC) - Endpoint (Week 8) | Week 8
  The WOMAC survey is used to assess joint-related discomfort at endpoint of the study. Our version of WOMAC score (adding up from all domains) can range from 0 (min) to 108 (max). The lower the number, the better the outcome (less joint-related discomfort).
The Visual Analog Scale (VAS) - Baseline | Baseline
  VAS is used for pain assessment at baseline. VAS ranges from 0 (min) to 10 (max). In our study, only those with VAS of 4 points or more at baseline were included, so our VAS ranges from 4 to 10, with the lower values indicating less pain, and thus better outcome.
The Visual Analog Scale (VAS) - Midpoint (Week 4) | Week 4
  VAS is used for pain assessment at midpoint. VAS ranges from 0 (min) to 10 (max). In our study, only those with VAS of 4 points or more at baseline were included, so our VAS ranges from 4 to 10, with the lower values indicating less pain, and thus better outcome.
The Visual Analog Scale (VAS) - Endpoint (Week 8) | Week 8
  VAS is used for pain assessment at endpoint. VAS ranges from 0 (min) to 10 (max). In our study, only those with VAS of 4 points or more at baseline were included, so our VAS ranges from 4 to 10, with the lower values indicating less pain, and thus better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rania Ibrahim, PhD, Principal Investigator — BioScreen Testing Services
Locations (1):
- Avicenna Nutraceutical, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No